CLINICAL TRIAL: NCT06152419
Title: Patient Education Videos to Improve Patients' Experience During Radiotherapy Treatment: a National Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Collaborators: Stichting tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONZ-2022-0579
Record Dates: First submitted 2023-11-06; First posted 2023-11-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Cancer, Breast; Cancer, Lung; Cancer Prostate; Cancer Head Neck; Cancer, Gastrointestinal
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: A first video illustrating the general radiotherapy process was created with voice-over in Dutch and French. The video will be shown to 125 patients undergoing radiotherapy in 3 Flemish and 2 Walloon radiotherapy departments. Patients will be asked to complete questionnaires to evaluate the quality and the impact of the video and to assess the need for additional information. Patients will be recruited at the first consultation at the radiotherapy department or at one of the first radiotherapy sessions. In addition, focus groups will be organised to assess whether this video meets the patients' needs. At least 25 patients at at UZ Gent will be invited to participate in 5 focus groups, each focus group concentrating on one of the 5 most frequent tumor groups. Based on the collected data, both a qualitative and quantitative. In a second phase, additional visual material will be created.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interrogated patients (Experimental): Patients will be asked to complete questionnaires to evaluate the quality and the impact of the video and to assess the need for additional information. Patients will be recruited at the first consultation at the radiotherapy department or at one of the first radiotherapy sessions. In addition, focus groups will be organised to assess whether this video meets the patients' needs.
  Interventions: Device: Questionnaire

INTERVENTIONS:
Device: Questionnaire — Patients will be asked to complete questionnaires to evaluate the quality and the impact of the video and to assess the need for additional information.

SUMMARY:
Patients often base their information on the experiences of other patients or on information they find on the internet. This information is in many cases incorrect, outdated or not applying to the patient's situation. This leads to misconceptions or inappropriate anxiety. During the intake consultation at the radiotherapy department, doctors, nurses and RTTs provide accurate and patient-specific information, but it can be overwhelming and it is known that only part of this information is remembered. Moreover, it remains difficult for a patient to imagine how the treatment will proceed.

The combination of verbal information, supplemented with video material, seems to be the ideal way to convey information. After all, a video can be viewed again afterwards, possibly together with loved ones, or can be shown in advance in preparation of the consultation. In Belgium, the existence of patient education videos about radiotherapy is very limited. Making these kinds of videos is expensive and time consuming. For that reason, BeSTRO (Belgian Society for Radiotherapy and Oncology) started a project to make videos for patients that can be used nationally by all radiotherapy centers. The project is sponsored by Foundation against Cancer.

DETAILED DESCRIPTION:
A first video illustrating the general radiotherapy process is already available. This video will be used as a 'test video' to be shown to patients undergoing radiotherapy in one of the 4 participating centers. Questionnaires will evaluate the quality and the impact of the video and will assess the need for additional information. Moreover, 25 patients will be invited to participate in 5 focus groups, each focus group concentrating on one of the 5 most frequent tumor groups (breast tumors, lung tumors, head and neck tumors, urological tumors and gastro-intestinal tumors). The information gathered from the questionnaires and focus groups will be used to determine the content and format of the next videos. In total, about 10 videos on specific parts of the radiotherapy process will be produced.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cancer,
* age ≥ 18 years,
* undergoing radiotherapy as part of their treatment

Exclusion Criteria:

- history of previous radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionaire to increase knowledge of radiotherapy | Trough study completion, an average of 1 year
  We will evaluate the patients' knowledge about radiotherapy using a questionnaire and various focus groups.The outcome measurement will be the personal opinion of the patient about his/her knowledge about radiotherapy (I feel more educated - the video has no value).
Patient questionnaire on radiotherapy-related anxiety | Trough study completion, an average of 1 year
  We will evaluate the patients' treatment-related-anxiety by providing additional information (by means of an educational video). The outcome measurement will be the personal opinion of the patient about his/her anxiety (less fear - equal fear - more fear).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitary Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No
The data of the questionnaires will be prospectively collected in the intelligent software database REDCap. Data collected include patient, tumour, diagnostic and treatment characteristics, and evaluation of the videos. The data is analyzed with statistical software.The group debate will be recorded. The recording will be destroyed after analysis of the data. The debate will be qualitatively processed with specific software, namely NVIVO.